CLINICAL TRIAL: NCT05468307
Title: A Clinical Study of Engineered Tumor Infiltrating Lymphocytes Injection (GC203 TIL) in Patients With Advanced Gynecologic Tumors
Brief Title: A Study of GC203 TIL in Advanced Gynecologic Tumors (10hospital)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC203-2022-10hospital-Gyne
Record Dates: First submitted 2022-06-16; First posted 2022-07-21 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2024-11

CONDITIONS: Advanced Gynecologic Tumors; TIL Engineered With Membrane-Binding Cytokine; Treatment Side Effects; Effects of Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Membrane Bound Cytokine Modified TIL (Experimental): 2x10^8-1x10^10 in vitro expanded autologous TIL engineered with membrane-binding cytokine (GC203 TIL) will be infused i.v. to patients with advanced gynecologic tumors after NMA lymphodepletion treatment with cyclophosphamide.
  Interventions: Biological: Membrane Bound Cytokine Modified TIL

INTERVENTIONS:
Biological: Membrane Bound Cytokine Modified TIL — Adoptive transfer of 2x10^8-1x10^10 autologous TIL engineered with membrane-binding cytokine to patients i.v. in 30-120 minutes.

SUMMARY:
This study is to investigate the safety and efficacy on TIL engineered with membrane-binding cytokine (GC203 TIL) for the treatment of patients with advanced gynecologic tumors. Autologous TILs from tumor resections or biopsies are first gene modified (engineered with membrane-binding cytokine) and than expanded before i.v. infusion into the patient after NMA lymphodepletion treatment with cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years to 75 years;
2. Histologically diagnosed as primary/relapsed/metastasized Gynecological tumors;
3. Expected life-span more than 3 months;
4. Karnofsky≥60% or ECOG score 0-2;
5. Test subjects have failed standard treatment regimens, or there are no standard treatment regimens available.
6. Test subjects must have tumor regions eligible for biopsy or resection, or malignant body fluid where TILs can be isolated;
7. At least 1 evaluable tumor lesion;
8. Hematology and Chemistry（within 7 days prior to enrollment）:

   * Absolute count of white blood cells≥2.5×10^9/L;
   * Absolute count of neutropils≥1.5×10^9/L;
   * Absolute count of lymphocytes ≥0.7×109/L；
   * Platelet count≥100×10^9；
   * hemoglobin≥90 g/L;
   * Activated partial thromboplastin time (APTT) ≤1.5xULN (Unless received anticoagulant therapy within the previous 3 days);
   * International normalized ratio (INR) ≤1.5xULN (Unless received anticoagulant therapy within the previous 3 days);
   * Serum creatinine ≤1.5mg/dL(or ≤132.6μmol/L), or clearance rate≥50mL/min;
   * Serum ALT/AST ≤3×ULN(subjects with liver metastasis ≤3×ULN);
   * Totol bilirubin≤1.5×ULN;
9. no absolute or relative contraindications to operation or biopsy;
10. Test subjects with child-bearing potential must be willing to practice approved highly effective methods of contraception at the time of informed consent, and continue within 1 year after the completion of lymphodepletion；
11. Any malignant tumor-targeting therapies, including radiotherapy, chemotherapy and biologics must cease 28 days before obtaining TILs;
12. Be able to understand and sign the informed consent document;
13. Be able to stick to follow-up visit plan and other requirements in the agreement.

Exclusion Criteria:

1. Need glucocorticoid treatment, and daily dose of Prednisone greater than 15mg (or equivalent doses of hormones) or outoimmune diseases requiring immunomodulatory treatment;
2. Forced expiratory volume in one second (FEV1) less than 2L, diffusing capacity of the lung for carbon monoxide (DLCO) (calibrated) less than 40%;
3. Significant cardiovascular anomalies according to any of the following definition: New York Heart Association (NYHA) Grade III or IV congestive heart failure, clinically significant low blood pressure, uncontrollable symptomatic coronary artery diseases, or ejection fraction less than 35%; Severe cardiac rhythm and conduction anomaly, such as ventricular arrhythmia requiring clinical intervention, second-third degree atrio-ventricular conductive block, etc.
4. Human immunodeficiency virus (HIV) infection or anti-HIV antibody positive, active HBV or HCV infection (HBsAg positive and/or anti-HCV positive), syphilis infection or Treponema pallidum antibody positive;
5. Severe physical or mental diseases;
6. Have a systemic active infection requiring treatment, or have positive blood cultures(or imaging evidence of infection);
7. Having been treated within a month or being treated now with other medicines, or other biologic therapy, chemo-or radiotherapy;
8. History of allergy to chemical compound consisting of chemical and biologic substances resembling cell therapy;
9. Having received immunotherapy and developed irAE level greater than Level 3;
10. Previous anti-tumor treatment AE did not return to CTCAE5.0 version grade 1 or below (toxicity considered by the investigator as non-safety concerns like alopecia excluded);
11. Females in pregnancy or lactation;
12. History of organ transplantation, allogeneic stem cell transplantation, and renal replacement therapy;
13. Researchers considering the test subject as having a history of other severe systemic diseases, or other reasons inappropriate for the clinical study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) | Up to 6 months
  To characterize the safety profile of TIL engineered with membrane-binding cytokine (GC203 TIL) in patients with advanced gynecologic tumors as assessed by incidence of adverse events related to GC203 TIL infusion.
Objective Response Rate (ORR) | Up to 36 months
  Proportion of patients with response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1):
  ORR (proportion of patients) = # with CR + # with PR / # with CR + # with PR + # with SD + # with PD.
  ( Except baseline evaluation within 28 days before GC203 TIL infusion，PET/CT scan will be performed at 6 weeks after GC203 TIL infusion, and than every 6 weeks for 6 months, and then every 6 months after that for up to 3 years)
Disease Control Rate (DCR） | Up to 36 months
  Percentage of patients that meet CR, PR and SD criteria set in this study according to RECIST v1.1： DCR (proportion of patients) = # with CR + # with PR + # with SD / # with CR + # with PR + # with SD + # with PD.
Duration of Response (DOR) | Up to 36 months
  The time length between the first confirmed objective response per RECIST 1.1 to the treatment and the subsequent disease progression per RECIST 1.1
Progression-Free Survival (PFS) | Up to 36 months
  The time length between GC203 TIL infusion and confirmed subsequent disease progression according to RECIST 1.1
Overall Survival (OS) | Up to 36 months
  The length of time from the date of the start of GC203 TIL treatment that the patients are still alive

SECONDARY OUTCOMES:
Change in Quality of Life | Up to 36 months
  Comparison of patients' quality of life before and after GC203 TIL treatment as assessed by the EORTC(The European Organization for Reasearch and Treatment of Cancer) QLQ-30(Quality of Life Questionnare-Core30 ) (V3.0). The outcome will be calculated by software from different dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China